CLINICAL TRIAL: NCT03578874
Title: A Combination of Sorafenib, Capecitabine and Oxaliplatin (SECOX) as Neoadjuvant Therapy in Patients With Locally Advanced Hepatocellular Carcinoma: A Phase II Study
Brief Title: SECOX as Neoadjuvant Therapy in Patients With Locally Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YAU Chung Cheung Thomas, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKU-MONC-HCC-003
Record Dates: First submitted 2018-05-20; First posted 2018-07-06 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SECOX (Experimental): Sorafenib 400 mg twice daily from Day 1 to 14, Capecitabine 850 mg/m2 twice daily from Day 1 to 7, Oxaliplatin 85 mg/m2 on Day 1
  Interventions: Drug: Sorafenib; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Sorafenib — PO
  Other Names: Nexavar
Drug: Capecitabine — PO
Drug: Oxaliplatin — IV

SUMMARY:
The purpose of this study is to evaluate the resectability after treatment with SECOX (sorafenib, capecitabine, oxaliplatin) as neoadjuvant therapy in patients with locally advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* HCC confined to single lobe of non-cirrhotic liver (locally advanced) and not suitable for surgery or loco-regional therapies at the time of study entry, but can become resectable after treatment
* Diagnosis of HCC confirmed by histology
* Child-Pugh class A cirrhosis with adequate remnant liver parenchyma
* Measurable disease
* Fit enough to undergo surgery to resect the primary liver tumour

Exclusion Criteria:

* Prior systemic therapy for HCC
* Presence of extrahepatic metastasis
* History of liver transplantation
* Peripheral sensory neuropathy with functional impairment
* Uncontrolled hypertension/ cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Resectability | At the end of Cycle 4 (each cycle is 14 days)
  Proportion of patients deemed resectable as assessed by designated hepatobiliary surgeons

SECONDARY OUTCOMES:
Objective response rate | At the end of Cycle 4 (each cycle is 14 days)
  Proportion of patients with a complete response (CR) or partial response (PR)
Progression-free survival | Approximately 18 months
  Time from study treatment to radiological disease progression or death due to any causes
Overall survival | Approximately 33 months
  Time from study treatment to the date of death due to any cause or last follow-up date

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong